CLINICAL TRIAL: NCT06953492
Title: Association Between Sleep State and Lung Cancer Prognosis: a Retrospective Study
Brief Title: Sleep State in Lung Cancer: A Retrospective Analysis
Status: Completed | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SD-lung cancer-Retrospective
Record Dates: First submitted 2025-04-16; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Lung Adenocarcinoma; Sleep Disorders, Circadian Rhythm
MeSH Terms: conditions — Adenocarcinoma of Lung; Sleep Disorders, Circadian Rhythm

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lung cancer: lung cancer-Non SD; lung cancer-SD
  Interventions: Other: PSQI

INTERVENTIONS:
Other: PSQI — PSQI

SUMMARY:
Lung cancer remains the leading cause of cancer-related mortality globally, with tumor progression closely linked to the immune microenvironment. Sleep disorders (e.g., insomnia, obstructive sleep apnea [OSA]) affect 40-50% of lung cancer patients and may promote tumorigenesis via chronic inflammation, immune suppression, and metabolic dysregulation. Preclinical and epidemiological studies suggest that chronic sleep deprivation reduces NK cell activity, elevates pro-inflammatory cytokines (IL-6, TNF-α), and upregulates angiogenic factors (VEGF), though clinical evidence remains scarce. This study aims to: Evaluate associations between sleep disorders and immunosuppressive phenotypes (e.g., PD-L1 expression, T-cell exhaustion) in lung cancer patients. Analyze the impact of sleep disturbances on immunotherapy efficacy (e.g., PD-1 inhibitors) and prognostic outcomes. Explore underlying mechanisms, including hypoxia-inducible factor (HIF-1α) signaling and sympathetic nervous system activation

DETAILED DESCRIPTION:
Lung cancer is the second most common cancer and the leading cause of cancer-related death in the world, and its treatment and prognosis improvement are still major clinical challenges. In recent years, tumor immunotherapy represented by immune checkpoint inhibitors has significantly improved the survival outcome of some patients, but the individual efficacy varies significantly, suggesting that tumor microenvironment (TME) and host factors (such as lifestyle and metabolic status) may affect the mechanism of immune response. In this context, sleep disorders, as a common accompanying symptom of cancer, have gradually become the focus of research.

The incidence of sleep disorders (such as insomnia and circadian rhythm disturbance) in patients with lung cancer is as high as 40%-70%. Sleep disorders often form symptom clusters with fatigue and pain, which significantly reduce the quality of life and treatment compliance of patients. Studies have shown that sleep disorders not only exacerbate inflammation through neuroendocrine pathways (such as increased cortisol level and inhibited melatonin secretion), but also are closely related to immunosuppression in the tumor microenvironment. For example, sleep deprivation can lead to increased levels of proinflammatory factors (such as IL-6 and TNF-α) in peripheral blood, and inhibit CD8+ T cell function and NK cell activity, thereby weakening the antitumor immune response.

Sleep affects tumor progression by regulating immune cell function and cytokine network. According to the study of the University of Tuebingen in Germany, complete sleep can enhance the activity of T cell integrin and enhance its killing ability against infected or cancerous cells. Sleep disorders can inhibit the function of immune cells and promote tumor immune escape by increasing stress hormones such as adrenaline. In addition, the association between sleep disorders and immunological indicators (such as imbalance of lymphocyte subsets and dynamic changes of PD-L1 expression) during chemotherapy or radiotherapy in lung cancer patients has been partially confirmed, suggesting that sleep disorders may be used as a biomarker to predict the efficacy of immunotherapy.

Although many studies have investigated the effect of sleep disorders on the immune function of cancer patients, the research on the mechanism of lung cancer still has the following shortcomings: (1) Most studies focus on the symptom management of sleep disorders, and lack of systematic analysis of the dynamic relationship between sleep disorders and tumor immune microenvironment; (2) The existing evidence is mostly based on small sample cross-sectional studies, and there is a lack of longitudinal data to support the causal association between sleep disorders and the efficacy of immunotherapy. (3) There is a lack of clinical translational research on whether sleep interventions (e.g., cognitive behavioral therapy, melatonin supplementation) can reverse immunosuppression and enhance treatment response.

Based on the above background, the aim of this study is to investigate the relationship between sleep disorders and lung cancer immune characteristics (such as PD-L1 expression, T cell infiltration) and prognosis of immunotherapy through retrospective analysis, and to provide theoretical basis for optimizing individualized treatment strategies. The results of this study are expected to promote the in-depth analysis of the "sleep-immune" regulatory mechanism, and lay the foundation for a new combined immune therapy integrating sleep management.

ELIGIBILITY:
Inclusion Criteria:

1. NSCLC or SCLC was diagnosed.
2. Patients have received immunotherapy (e.g., PD-1/PD-L1 inhibitors) or standard treatment (chemotherapy/radiotherapy).
3. Sleep disorder diagnoses and immune-related biomarkers fully recorded in medical records.

Exclusion Criteria:

1. The patient had a history of other malignant tumors.
2. Key clinical data lacking.
3. The presence of a serious psychiatric or neurologic condition.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Data source and time range Data source: Adult patients (≥18 years old) diagnosed with primary lung cancer (confirmed by histopathology) in [Zhong Shan Hospital] from January 2018 to January 2025 were retrospectively enrolled.
  Data extraction: Clinical, pathological and follow-up data were collected through the electronic medical record system (EMR) and the hospital cancer registry database.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
OS | Baseline
  Overall survival (OS) : time from immunotherapy initiation to all-cause death

CONTACTS AND LOCATIONS:
Locations (1):
- Zhong Shan hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No